CLINICAL TRIAL: NCT02237313
Title: Identification of Vulnerability Factors in the Course of Pemphigus Patients - SHS Pemphigus Clinical Trial
Brief Title: Identification of Vulnerability Factors in the Course of Pemphigus Patients
Acronym: SHS-Pemphigus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Other
Other Study IDs: 2014/063/HP; 2014A0067740 (Registry Identifier: RCB number)
Record Dates: First submitted 2014-09-01; First posted 2014-09-11 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pemphigus; Dermatological Disease
Keywords: psychological support; therapeutic education; vulnerability of patients
MeSH Terms: conditions — Pemphigus; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- prevalent cases (Experimental): 40 prevalent cases correspond to patients with known pemphigus. Emphasis will be on included patients at different times of the course of their disease.
  8 incident cases recruited through the center of Rouen and following an intervention program with psychological support and therapeutic education program
  Interventions: Behavioral: psychological support and therapeutic education program

INTERVENTIONS:
Behavioral: psychological support and therapeutic education program

SUMMARY:
The bullous pemphigoid treatment is based on corticosteroids continued for several years. Pemphigus causes some patients a psychological impact and sometimes major vulnerability that can occur not only at diagnosis but also at later stages of disease progression. Our hypothesis is that these episodes of vulnerability may be under four kinds of factors that may be connected to the plurality of the history of these patients, and the resources they can mobilize throughout this experience, generating inequality in management and "work" around the disease.

DETAILED DESCRIPTION:
The originality of the project lies in its multidisciplinary approach (dermatology, psychology, sociology). No such study has yet been carried out in the pemphigus who has been the subject of a very small number of works in sociology or psychology. The only studies are studies of quality of life with no longitudinal follow-up. The perspective of qualitative and quantitative data, sociological and psychological approaches, should allow more innovative and adapted to the medico-social and psychological care of patients with pemphigus approaches. The purpose of this study is to identify the determinants leading to moments of vulnerability in the course of patients with pemphigus in order to be able to offer preventive or corrective actions to improve the experience of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient major
* Patients with pemphigus vulgaris, diagnosed on a combination of:

  1. clinical signs and
  2. histological image above basal epithelial detachment with intra acantholysis,
  3. direct immunofluorescence showing deposition of Immunoglobulin G and / or C3 to the surface of keratinocytes
* Join a social security scheme
* patient has been informed and have signed consent to participate in the study

Exclusion Criteria:

* Person placed under judicial protection,
* Patient without liberty by administrative or judicial decision,
* Patient participating in another trial for the duration of monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
analysis of vulnerability factors | 12 months
  evaluation of : perception by the patient of misdiagnosis, perception of a possible difference in assessment of the severity of his illness between himself and healthcare professionals, patient behavior in relation to available information sources, and the influence of information gathered on the illness experience, Patient trajectory during the diagnostic phase using individual interview and questionnaire

SECONDARY OUTCOMES:
analysis of vulnerability factors | 6 months
  evaluation of : perception by the patient of misdiagnosis, perception of a possible difference in assessment of the severity of his illness between himself and healthcare professionals, patient behavior in relation to available information sources, and the influence of information gathered on the illness experience, Patient trajectory during the diagnostic phase using individual interview and questionnaire
assessment of anxiety, uncertainty, fear, coping strategies | 12 months
  assessment of anxiety, uncertainty, fear, coping strategies using individual interview and questionnaire
assessment of anxiety, uncertainty, fear, coping strategies | 6 months
  assessment of anxiety, uncertainty, fear, coping strategies using individual interview and questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Joly, Professor, Principal Investigator — University Hospital, Rouen
Locations (9):
- France (9):
  - Hôpital Avicenne, Bobigny
  - CHU de Clermont-Ferrand Hôpital d'Estaing, Clermont-Ferrand
  - CH du Mans, Le Mans
  - CHRU de Lille Hôpital Claude Huriez, Lille
  - Hôpital La Timone, Assistance publique hôpitaux de Marseille-Aix, Marseille
  - Hôpital Haut-Lévêque, Pessac
  - Centre hospitalier de Cornouaille, Quimper
  - Hôpital Robert Debré, chu de Reims, Reims
  - University Hospital of Rouen, Rouen